CLINICAL TRIAL: NCT05662436
Title: Protocol for the Open Sky School: A Two-arm Clustered Randomized Controlled Trial to Test the Effectiveness of a Nature-based Intervention on Mental Health of Elementary School Children
Brief Title: Protocol for the Open Sky School
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McGill University (Other)
Collaborators: Observatory for Children's Education and Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 468540
Record Dates: First submitted 2022-11-25; First posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Child Behavior
Keywords: school-based intervention; mental health; children; randomized controlled trial; nature; outdoor education; elementary-school children; greenspace
MeSH Terms: conditions — Child Behavior; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The exposure to nature consists of teachers bringing their students to the highest quality green space within 1 km of a school which could be located on or off campus. The class will spend a total of 2 hours (i.e. 2 one hour visits or one 2 hours visits) per week for 12 weeks (transportation included). The teacher be provided with a toolkit of activities (mental health and academic competencies) that they will carry out with their students. Teachers will be provided with training and support.
  Interventions: Other: Open Sky School program
- Control (No Intervention): Six months after the inception of the trial, elementary schools (and their teachers) in the control condition will receive an unguided version of the intervention, supplemented by an online peer support group. As the children of the control group will by then be in high school with different teachers, we will provide them with a toolkit of 10 mental health activities that they can practice alone, in addition of support via video-conference, phone or email if they require help practicing the activities from a member of the research team. As in the intervention group, we will provide support by licensed psychologists to any children who report high levels of psychological distress and orient children to appropriate services if needed.

INTERVENTIONS:
Other: Open Sky School program — Teachers lead students in 2 hours of outdoor activities per week for 12 weeks, as detailed in the arm description
  Arms: Intervention group

SUMMARY:
The goal of this a randomized controlled trial to test the effectiveness of a nature-based intervention called Open Sky School to reduce mental health problems among elementary school children. More specifically a two-arm clustered randomized controlled trial will be conducted in elementary schools across Québec, Canada. Following informed consent by teachers, parents and students, schools will be randomly assigned 1:1 to the intervention or the control group with a total of 2500 6th grade students and 100 teachers expected to participate. The primary and secondary research questions are as follows.

The primary research question :

* Is the intervention effective in reducing mental health problems in children from pre-to-post test (Social Behavior Questionnaire: self and teacher reports) ?

The secondary research questions:

* Is the intervention effective in improving children's depression, positive and negative affect, nature connectedness. eco-anxiety and pro-environmental behaviors ?
* Is the intervention effective in improving teachers' well-being and affect ?
* Are the benefits to children sustained benefits at 3 months follow-up ?
* Is the primary question moderated by child's sex, child's disability status, the green space of neighbourhoods, the school's socio-economic position and teacher's experience wtih outdoor education ?

The intervention will take place outdoors in a green-space (2 hours per week for 12 weeks) and include a toolkit of 30 activities to foster well-being (e.g. mindfulness) and academic competencies (e.g. mathematics). The control group will engage in teaching-as-usual and will be provided with the activity toolkit after the trial has been conducted. Questionnaires will be administered to students before, immediately after and 3 months after the intervention in both the control and intervention groups. Teachers in both groups will complete questionnaires before and immediately after the intervention.

ELIGIBILITY:
Additional inclusion criteria for schools are: (a) access to a natural environment (e.g., park, wooden area) on school grounds or within 1 km of the school and (b) having 6th grade teachers provide informed and written consent to participate in this study. Inclusion criteria for children are (a) enrollment in 6th grade, (b) providing their assent and (c) having their parents or legal guardians provide informed written consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2022-12-20 (Estimated); Primary Completion 2023-06-20 (Estimated); Study Completion 2023-09-23 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Child Mental Health at 3 months | Baseline, 3 months
  The Social Behavior Questionnaire is a 30 items questionnaire that will be used to assess a range of mental health symptoms in children. The frequency of children's symptoms over the last 2 months is rated on a scale 3-point (never/not true = 0, sometimes/somewhat true = 1, often/very true = 2). Overall symptoms will be examined as outcomes, as well as internalizing symptoms (emotional distress and withdrawal; 11 items), externalizing symptoms (impulsive/hyperactive/inattentive and disruptive behaviors; 13 items), and social behaviors (pro-social behavior and peer relationships; 6 items). Ratings will be obtained by both child and teacher reports which will be analyzed separately.

SECONDARY OUTCOMES:
Change from Baseline Child Mental Health at 6 months | Baseline, 6 months
  The Social Behavior Questionnaire is a 30 items questionnaire that will be used to assess a range of mental health symptoms in children. The frequency of children's symptoms over the last 2 months is rated on a scale 3-point (never/not true = 0, sometimes/somewhat true = 1, often/very true = 2). Overall symptoms will be examined as outcomes, as well as internalizing symptoms (emotional distress and withdrawal; 11 items), externalizing symptoms (impulsive/hyperactive/inattentive and disruptive behaviors; 13 items), and social behaviors (pro-social behavior and peer relationships; 6 items). Ratings will be obtained the child self report version.
Change from Baseline Child Depressive symptoms at 3 months | Baseline, 3 months
  The Children's Depression Inventory-Short Version (CDI-S) includes 13 items that will be used to assess cognitive, affective and behavioral signs of depression in children. The CDI-S has good convergent, discriminate and factorial validity among children. Children consider how they were feeling over the last 2 weeks and respond on a 3-point scale (e.g. 1=I hate myself; 2=I don't like myself; 3=I like myself).
Change from Baseline Child Depressive Symptoms at 6 months | Baseline, 6 months
  The Children's Depression Inventory-Short Version (CDI-S) includes 13 items that will be used to assess cognitive, affective and behavioral signs of depression in children. The CDI-S has good convergent, discriminate and factorial validity among children. Children consider how they were feeling over the last 2 weeks and respond on a 3-point scale (e.g. 1=I hate myself; 2=I don't like myself; 3=I like myself).
Change from Baseline Child Positive and Negative Affect at 3 months | Baseline, 3 months
  The Positive and Negative Affect Schedule for Child (PANAS-C) is a 20-item scale that will be used to assess positive (e.g., "excited") and negative (e.g., "upset") affect which has good convergent and discriminate validity among children. Children will indicate to what extent they feel over the last weeks (1=very slightly or not at all; 5=extremely).
Change from Baseline Child Positive and Negative Affect at 6 months | Baseline, 6 months
  The Positive and Negative Affect Schedule for Child (PANAS-C) is a 20-item scale that will be used to assess positive (e.g., "excited") and negative (e.g., "upset") affect which has good convergent and discriminate validity among children. Children will indicate to what extent they feel over the last weeks (1=very slightly or not at all; 5=extremely).
Change from Baseline Child Connection with Nature at 3 Months | Baseline, 3 months
  The Nature Connection Index (NCI) is a self-report questionnaire including 6 items that will be used to assess connectedness to nature. The scale has good validity and reliability among children. Participants respond to affirmations (e.g. nature always makes me happy) using a 7-point scale (1=strongly agree; 7=strongly disagree).
Change from Baseline Child Connection with Nature at 6 Months | Baseline, 6 months
  The Nature Connection Index (NCI) is a self-report questionnaire including 6 items that will be used to assess connectedness to nature. The scale has good validity and reliability among children. Participants respond to affirmations (e.g. nature always makes me happy) using a 7-point scale (1=strongly agree; 7=strongly disagree).
Change from Baseline Child Pro-environmental Behaviors at 3 Months | Baseline, 3 months
  Pro-environmental attitude and behaviors will be measured with two questionnaires. The first is a brief 6-item measure developed in a recent study, asking children to report the frequency they made an effort to conserve water, energy and recycle trash (1=always; 5=never) and the extent to which they agree that they are ready to volunteer, give money and talk to their entourage to protect nature (1=strongly agree; 4=strongly disagree). The second includes 4 questions specific to climate change which were adapted from a previous study and developed by experts in the field. Children report the extent to which they are worried about climate change (1=not at all worried; 4=extremely worried), that these worries motivate them to engage in pro-environmental behaviors or activism (1=not at all; 4=a lot) and that they feel capable of making behavioral changes to help the environment (1=strongly disagree; 4=strongly agree).
Change from Baseline Child Pro-environmental Behaviors at 6 Months | Baseline, 6 months
  Pro-environmental attitude and behaviors will be measured with two questionnaires. The first is a brief 6-item measure developed in a recent study, asking children to report the frequency they made an effort to conserve water, energy and recycle trash (1=always; 5=never) and the extent to which they agree that they are ready to volunteer, give money and talk to their entourage to protect nature (1=strongly agree; 4=strongly disagree). The second includes 4 questions specific to climate change which were adapted from a previous study and developed by experts in the field. Children report the extent to which they are worried about climate change (1=not at all worried; 4=extremely worried), that these worries motivate them to engage in pro-environmental behaviors or activism (1=not at all; 4=a lot) and that they feel capable of making behavioral changes to help the environment (1=strongly disagree; 4=strongly agree).
Child's Appreciation of the Program | 3 months
  We designed one item for children to self-report the frequency that they appreciated the intervention (1=not at all; 4=always) that will be administered in the intervention group at post-test.
Change from Baseline Teacher Well-being at 3 Months | Baseline, 3 months
  The World Health Organization Well-Being Index (WHO-5) is a 5-item self-report measure that will assess of wellbeing for adults. The WHO-5 is a widely used, valid and reliable measure that is sensitive to change. Participants indicate the frequency of their feelings (e.g. in a good mood) over the last two weeks (5=all the time; 0=never).
Change from Baseline Teacher Positive and Negative Affect at 3 Months | Baseline, 3 Months
  The Positive and Negative Affect Schedule (PANAS) is a 20-item scale that will be used to assess positive (e.g., "excited") and negative (e.g., "upset") affect which has well-established good psychometric properties. Teachers will indicate to what extent they feel over the last weeks (1=very slightly or not at all; 5=extremely).
Teacher's Enjoyment of Outdoor Education | 3 months
  An adapted version of the Enjoyment of Teaching Mathematics Scale will be used for teachers from the intervention group at post-test to self-report their enjoyment of teaching outdoors (e.g. I really like teaching outdoors) with 5 items on a 5 point scale (1=strongly agree; 5=strongly disagree).
Teacher's Qualifications and Experience | Baseline
  We designed questions about teachers qualification and experience teaching in general. Higher scores indicate higher levels of experience.
  This will be investigated as a moderator.
Teacher's Experience Teaching Outdoors | Baseline
  Teachers' experience with outdoor teaching over the last 3 years (e.g. context, duration) (e.g. did you practice outdoor education in autumn 2022?) and outdoor activities practiced in their leisure time will be assessed with a 6 questions that were successfully used in a previous study on school based outdoor education. Higher scores indicate higher levels of experience outdoors. This will be investigated as a moderator.
Green Space of Neighborhoods | Baseline
  The Normalized Difference Vegetation Index (NDVI) will be used to quantify the density of green vegetation associated with the school's zip code. The widely used NDVI is based on the land surface reflectance of colors which is drawn from satellite images of the earth's surface. The index varies between +1 and -1 with higher values indicating higher green vegetation density. We will use 2019 satellite images which are available via the Consortium CANUE. This will be investigated as a moderator.
Disability Status of Children | Baseline
  Children formally diagnosed as having a physical or mental disability (e.g. intellectual deficiency) or having adaptation disorders (e.g. conduct disorders) or learning disorders (e.g. language deficits) will be identified via their school records. This will be investigated as a moderator.
Child's Sex | Baseline
  The children's sex (male, female) will be obtained via school records. This will be investigated as a moderator.
School's Level of Socio-economic Deprivation | Baseline
  School's level of deprivation will be quantified using a ranking provided by the Ministry of Education and Higher Education. The ranking is based on a composite score incorporating the proportion of students within each school whose mother completed high-school and whose both parents are employed full time. Schools are classified on a scale ranging from 1 (lowest deprivation) to 10 (highest deprivation) and scores of 8 to 10 are considered as disadvantaged. This will be investigated as a moderator

OTHER OUTCOMES:
Adherence Assessments: Teacher Logbook | Weekly during the intervention phase (12 weeks) in the intervention group
  The teachers will keep a logbook in which they will indicate information about each nature visit. They will provide information on the activities they chose to carry out (from our toolkit or others of their choice), the duration of these activities, where the activity was carried out and the total time spent outdoors. They will record if they watched our training videos, if they encountered any problems and the amount of time they spent with our supervisors. This information will be used to evaluate the adequacy of the implementation of our intervention. To fully comply with implementation, there must be of a total of 24 hours of intervention (2 hours per week for 12 weeks) and a minimum of 10 mental health activities from the toolkit must be carried out.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Claude Geoffroy, PhD, Principal Investigator — McGill
Locations (1):
- Douglas Mental Health University Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Loose T, Fuoco J, Malboeuf-Hurtubise C, Ayotte-Beaudet JP, Gauvin L, Chadi N, Ouellet-Morin I, Masse B, Cote SM, Geoffroy MC. A Nature-Based Intervention and Mental Health of Schoolchildren: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2024 Nov 4;7(11):e2444824. doi: 10.1001/jamanetworkopen.2024.44824. PMID 39546315
- [Derived] Loose T, Cote S, Malboeuf-Hurtubise C, Beaudet JA, Lessard G, Chadi N, Gauvin L, Morin IO, Geoffroy MC. Protocol for the Open Sky School: a two-arm clustered randomized controlled trial to test the effectiveness of a nature-based intervention on mental health of elementary school children. BMC Public Health. 2023 Feb 3;23(1):236. doi: 10.1186/s12889-023-15033-y. PMID 36737725